CLINICAL TRIAL: NCT02073864
Title: Neurological Complications of Contemporary Unprotected TAVR (Yale Neuro TAVR)
Brief Title: A Study to Evaluate the Neuro-embolic Consequences of TAVR
Status: Completed | Type: Observational
Sponsor: Keystone Heart (Industry)
Responsible Party: Sponsor
Other Study IDs: Yale Neuro TAVR
Record Dates: First submitted 2014-02-23; First posted 2014-02-27 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Aortic Valve Stenosis
Keywords: Aortic valve stenosis, stenosis, intervention
MeSH Terms: conditions — Aortic Valve Stenosis; Constriction, Pathologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A prospective, multi-center study to evaluate the neuro-embolic consequences of Transcatheter Aortic Valve Replacement (TAVR)

DETAILED DESCRIPTION:
Prospective, multi-center study enrolling a minimum of 20 up to a maximum of 80 patients at up to six investigational sites in the United States and European Union. Patients meeting eligibility criteria for TAVR will be enrolled to undergo diffusion-weighted MRI brain imaging pre-procedure (optional) and post-procedure and neuropsychological testing pre- and post-procedure, and at 30 days of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be ≥18 years of age.
* Patient meets indications for TAVR procedure.
* The patient is willing to comply with protocol-specified follow-up evaluations.
* The patient, or legally authorized representative, has been informed of the nature of the study, agrees to its provisions and has provided written informed consent, approved by the appropriate Institutional Review Board (IRB) or Ethics Committee (EC).

Exclusion Criteria:

* Patients undergoing TAVR via the trans-axillary, subclavian, or direct aortic route
* Pregnant or nursing subjects and those who plan pregnancy in the period up to 1 year following index procedure. Female subjects of child-bearing potential must have a negative pregnancy test done within 7 days prior to index procedure per site standard test.
* Patients with known diagnosis of acute myocardial infarction (AMI) within 72 hours preceding the index procedure (according to definition) or AMI >72 hours preceding the index procedure, in whom creatine kinase and creatine kinase have not returned to within normal limits at the time of procedure.
* Patients who are currently experiencing clinical symptoms consistent with new onset AMI, such as nitrate-unresponsive prolonged chest pain.
* Patients with impaired renal function (estimated Glomerular Filtration Rate [Estimated Glomerular Filtration Rate] <30, calculated from serum creatinine by the Cockcroft-Gault formula).
* Patients with a platelet count of <100.000 cells/mm³ or > 700.000 cells/mm³ or a white blood cell< 3000 cells/mm³ within 7 days prior to index procedure or per standard local practice.
* Patients with a history of bleeding diathesis or coagulopathy or patients in whom anti-platelet and/or anticoagulant therapy is contraindicated, or who will refuse transfusion.
* Patients who have received any organ transplant or are on a waiting list for any organ transplant.
* Patients with known other medical illness or known history of substance abuse that may cause non-compliance with the protocol, confound the data interpretation or is associated with a life expectancy of less than one year.
* Patients with known hypersensitivity or contraindication to aspirin, heparin/bivalirudin, clopidogrel/ticlopidine, nitinol, stainless steel alloy, and/or contrast sensitivity that cannot be adequately pre-medicated.
* Patients with a history of a stroke or transient ischemic attack (TIA) within the prior 6 months.
* Patients with an active peptic ulcer or history of upper gastrointestinal (GI) bleeding within the prior 6 months.
* Patients presenting with cardiogenic shock.
* Patients with documented friable or mobile atherosclerotic plaque in the aortic arch.
* Patients with contraindication to cerebral MRI.
* Patients with any other cardiovascular procedure prior to TAVR
* Patients with severe aortic arch atheroma visible on CT scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients indicated for TAVR procedure
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2013-11; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Incidence of diffusion-weighted MRI lesions following TAVR without cerebral embolic protection | 1 week post procedure
  Number of new diffusion-weighted MRI lesions

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Lansky, Md., Principal Investigator — Yale Cardiovascular Clinical Research
Locations (5):
- United States (5):
  - Yale New Haven Hospital, New Haven, Connecticut
  - Baptist Hospital of Miami, Miami, Florida
  - Columbia University Medical Center, Fort Lee, New Jersey
  - St. Francis Hospital, Roslyn, New York
  - The Heart Hospital Baylor Plano, Plano, Texas